CLINICAL TRIAL: NCT00658476
Title: Treating Adolescent Depression With Fish Oils
Brief Title: Omega-3 Fatty Acids for Treatment of Depression in Adolescents
Acronym: PUFA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Dr. Sayed Naqvi, M.D., Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9407
Record Dates: First submitted 2008-04-08; First posted 2008-04-15 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Adolescent Depression; Depression; Teenage Depression; Los Angeles
MeSH Terms: conditions — Depression | interventions — Fish Oils; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Fatty Acids (Experimental): Adolescents receive cognitive behavior therapy in combination with Omega-3 fatty acid supplements.
  Interventions: Dietary Supplement: Fish Oil; Behavioral: Cognitive Behavior Therapy
- Placebo (Placebo Comparator): Adolescents receive cognitive behavior therapy in combination with placebo.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — Omega-3 fatty acid supplements.
  Arms: Omega-3 Fatty Acids
Behavioral: Cognitive Behavior Therapy — Adolescents receive cognitive behavior therapy.
Other: Placebo
  Arms: Placebo

SUMMARY:
Adolescence is the highest risk period for depression onset. More than 1.3 million youths suffer from major depression annually in the United States, and there is evidence for an increasing trend. Because many adolescents have their first depressive episode in adolescence and adolescent depression often leads to recurrent mood disorders in adults, effective treatment during early illness can minimize the negative consequences of initial and repeated episodes. Although some antidepressants (particularly Selective serotonin reuptake inhibitors (SSRIs)) are effective treatments for juvenile depression, recent warnings about suicide and the use of SSRls highlight the need for new and safe treatment for juvenile depression. Data in adults suggest that supplementation with polyunsaturated fatty acids (PUFA) might be useful for the treatment of depression. The purpose of this study is to investigate the safety and efficacy of PUFA for the treatment of adolescent depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents between the ages of 13 and 21 currently under standard of care treatment at the Child Division of the Department of Psychiatry at CSMC
2. Diagnosed with major depressive disorder using the DSM-IV diagnostic criteria

Exclusion Criteria:

1. Active suicidal ideation, with a current plan and/ or a recent suicide attempt
2. Severe psychotic symptoms (presence of distressing or common hallucinations and/ or delusions)
3. History of bipolar disorder, eating disorder, schizophrenia, schizoaffective disorder, or autism
4. Potential subjects using psychotropic medication(s), alcohol, and/ or drugs within 2 weeks prior to entry into the study (8 weeks for fluoxetine and MAOIs - monoamine oxidase inhibitors)
5. Pregnant or lactating females, or those who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy) and become pregnant
6. Seizure or other neurological disorders
7. Dermatological conditions
8. Unstable cardiac, pulmonary, endocrine, or renal disorder
9. Adolescents who are currently being effectively treated with antidepressants

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Child Depression Inventory - CDI | 8 times for an average of 8 weeks
Hamilton Depression Rating Scale | 8 times for an average of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Naqvi, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States